CLINICAL TRIAL: NCT03139487
Title: A Randomized Phase II Open Label Study to Compare the Safety and Efficacy of Subcutaneous Dalteparin Versus Direct Oral Anticoagulants for Cancer-associated Venous Thromboembolism in Patients With Advanced Upper Gastrointestinal, Hepatobiliary and Pancreatic Cancer: PRIORITY
Brief Title: A Randomized Phase II Open Label Study to Compare the Safety and Efficacy of Subcutaneous Dalteparin Versus Direct Oral Anticoagulants for Cancer-associated Venous Thromboembolism
Acronym: PRIORITY
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sook Ryun Park, Associated professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2017-0327
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Cancer-associated Thrombosis; Esophageal Cancer; Stomach Cancer; Hepatocellular Carcinoma; Pancreatic Cancer; Duodenal Cancer; Esophagogastric Junction Cancer; Malignant Gastrointestinal Stromal Tumor; Ampulla of Vater Cancer; Biliary Cancer (Cholangiocarcinoma, Gall Bladder Cancer)
Keywords: Anticoagulant Adverse Reaction; Cancer-associated Thrombosis; Low molecular weight heparin; Direct oral anticoagulant
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Carcinoma, Hepatocellular; Pancreatic Neoplasms; Duodenal Neoplasms; Gastrointestinal Stromal Tumors; Biliary Tract Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms | interventions — Rivaroxaban; Dalteparin; apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Low molecular weight heparin (Active Comparator): Dalteparin, 200 IU/kg subcutaneously once daily for 4 weeks followed by 150 IU/kg once daily for 20 weeks
  Interventions: Drug: Dalteparin
- Direct oral anticoagulant (Experimental): Rivaroxaban, 15 mg orally twice daily for 3 weeks followed by 20mg once daily for 21 weeks
  Apixaban, 10 mg orally twice daily for 7days followed by 5mg twice daily for 21 weeks
  Interventions: Drug: Rivaroxaban; Drug: apixaban

INTERVENTIONS:
Drug: Rivaroxaban — 15 mg q12 hours for 3 weeks followed by 20mg q24 hours for 21 weeks
  Other Names: Xarelto
  Arms: Direct oral anticoagulant
Drug: Dalteparin — 200 IU/kg q24 hours for 4 weeks followed by 150 IU/kg q24 hours for 20 weeks
  Other Names: Fragmin
  Arms: Low molecular weight heparin
Drug: apixaban — 10 mg q12 hours for 7days followed by 5mg q12 hours for 21 weeks
  Other Names: eliquis
  Arms: Direct oral anticoagulant

SUMMARY:
This is an open label, multi-center, and randomized phase II trial designed to compare the safety and efficacy of direct oral anticoagulants and subcutaneous dalteparin in patients with acute venous thromboembolism and upper gastrointestinal, hepatobiliary, or pancreatic cancer, based on a group sequential design. Enrolled patients will be randomized in a 1:1 ratio. Patients will be stratified by performance status, type of cancer, chemotherapy and medical centers.

DETAILED DESCRIPTION:
This randomized II clinical trial will enrol patients with advanced upper gastrointestinal, hepatobiliary and pancreatic cancer who have venous thromboembolism (VTE), including pulmonary embolism and deep vein thrombosis. Patients will be randomized in a 1:1 ratio and stratified by performance status, type of cancer and medical centers. The enrolled patients will receive either subcutaneous dalteparin or DOAC(rivaroxaban, apixavan) according to randomization until the end of planned treatment schedules (six months), recurrence of VTE, clinical relevant bleeding, major bleeding, death or discontinuation of study treatment for any other reason (e.g. withdrawal of consent or discretion of the investigator). The primary end-point is the rate of clinical relevant bleeding event as defined as overt bleeding which was associated with medical intervention. In addition to time to clinical relevant bleeding event, time to event of major bleeding, total bleeding including minor event, time to recurrent VTE, overall bleeding rate and overall VTE recurrent rate will be analyzed to compare safety and efficacy of both anticoagulants. The final analysis will be conducted when the last enrolled patient has an event or has completed as least six months follow up in the study. Patients without bleeding and recurrent VTE events at data cut-off are censored at the last date the patient is known to be free of events.

Planned interim analysis will be conducted in the intentions to treatment analysis set. The interim analysis for the randomized portion of the study will be performed when at least 40% of estimated bleeding events have been observed. The purpose of interim analysis is for early stopping of the study for safety. This study will use a Data Monitoring Committee.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic active cancer including Esophageal cancer, Esophagogastric junction cancer, Stomach cancer, Gastrointestinal stromal disease, Ampulla of Vater cancer, Duodenal cancer, Hepatocelluar carcinoma, Biliary cancer (cholangiocarcinoma, gall bladder cancer), Pancreatic cancer
* Newly diagnosed deep vein thrombosis in any site and/or pulmonary thromboembolism on the basis of CT or doppler ultrasound image with or without symptoms
* Male or female ≥ 18 years, < 80 years old age
* Adequate major organ function including the following: Hematopoietic function: Platelet ≥ 75,000/mm3, Hepatic function: alanine aminotransferase levels 3 x upper limit of normal (if, with liver metastasis, alanine aminotransferase levels 5 x upper limit of normal), Aspartate Transaminase levels 3 x upper limit of normal (if, with liver metastasis, Aspartate Transaminase levels 5 x upper limit of normal), Renal function: estimated glomerular filtration rate ≥ 30 ml/min, Adequate coagulation time: prothrombin time ≤ 2 international normalized ratio, activated partial thromboplastin time 1.5 x upper limit of normal
* Able to understand and comply with the requirement of the study and to provide written informed consent

Exclusion Criteria:

Patients will be excluded from the study for any of the following reasons:

* Hemodynamically unstable pulmonary thromboembolism
* Use with P-gp and strong CYP3A4 Inhibitors (e.g., ketoconazole, itraconazole, lopinavir/ritonavir, ritonavir, indinavir/ritonavir, and conivaptan) or inducers (e.g., carbamazepine, phenytoin, rifampin, St. John's wort)
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome (e.g. patients with partial or total gastrectomy can enter the study, but not those with a jejunostomy probe), or inability to take oral medication
* Patients with current bleeding
* Recent history of major or uncontrolled bleeding within the previous 4 weeks
* Severe malnutrition, BMI < 16
* Patients who are receiving a therapeutic dose of rivaroxaban, low molecular weight heparin, fondaparinux, or unfractionated heparin for more than 72 hours before enrollment
* Administration of a fibrinolytic agent for treatment of the current episode
* Uncontrolled systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg
* Patients who have to keep concurrent antiplatelet agent (e.g. aspirin, clopidogrel)
* Patients who have clinical significant liver cirrhosis (Child Pugh score ≥ 7)
* Inadequate cardiovascular function: New York Heart Association class III or IV heart disease, Unstable angina or myocardial infarction within the past 6 months, History of significant ventricular arrhythmia requiring medication with antiarrhythmics or significant conduction system abnormality
* Serious concurrent infection or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy, including infective endocarditis
* History of or current brain metastases
* Life expectancy less than 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2017-08-07 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of clinical relevant bleeding | 6 months
  Clinically relevant bleeding: overt bleeding which was associated with medical intervention, unscheduled contact with a physician, interruption or discontinuation of anticoagulation, or associated with any other discomfort such as pain or impairment of activities of daily life, including major bleeding

SECONDARY OUTCOMES:
Rate of major bleeding | 6 months
  Major bleeding: Contributing to death, associated with a fall in hemoglobin ≧ 2 g/dL, or leading to transfusion of ≧ 2 units of red cells or if bleeding is intracranial, retroperitoneal, or another critical site.
Rate of total event of bleeding | 6 months
Time to major bleeding event | 6 months
Time to clinical relevant bleeding event | 6 months
Time to total event of bleeding | 6 months
Rate of recurrent or aggravated venous thromboembolism | 6 months
Time to recurrent or aggravated venous thromboembolism | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riaz IB, Fuentes HE, Naqvi SAA, He H, Sipra QR, Tafur AJ, Padranos L, Wysokinski WE, Marshall AL, Vandvik PO, Montori V, Bryce AH, Liu H, Badgett RG, Murad MH, McBane RD 2nd. Direct Oral Anticoagulants Compared With Dalteparin for Treatment of Cancer-Associated Thrombosis: A Living, Interactive Systematic Review and Network Meta-analysis. Mayo Clin Proc. 2022 Feb;97(2):308-324. doi: 10.1016/j.mayocp.2020.10.041. Epub 2021 Jun 22. PMID 34172290